CLINICAL TRIAL: NCT01064531
Title: A Randomized Controlled Trial to Compare Implant Migration of the MIS Stem Versus The Synergy Total Hip System by Radiostereometric Analysis
Brief Title: Mini Stem Radiostereometric Analysis Study
Acronym: MISRSA
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: US-CR-130
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- MIS Femoral Neck Stem: Subject will be randomized to either MIS or Synergy implant.
  Interventions: Device: MIS Femoral Neck Stem implant
- Synergy Hip System: Subject will be randomized to either Synergy or MIS implant.
  Interventions: Device: MIS Femoral Neck Stem implant

INTERVENTIONS:
Device: MIS Femoral Neck Stem implant

SUMMARY:
The objectives of this study are to assess migration of the MIS Stem compared to the Synergy Hip System using Radiostereometric Analysis (RSA), and to assess the long-term safety and effectiveness of the study device. This study will document any device-related surgical or post-operative complications and adverse radiographic observations.

Subjects meeting the entrance criteria specified in this protocol will be randomized as they become available.

DETAILED DESCRIPTION:
The purpose of the current investigation is to compare migration of the device after implantation with a modular, short hip stem called the "MIS Stem" or a standard THA using the Synergy Hip System using RSA. The intended use of this product is for patients with inflammatory and non-inflammatory degenerative joint disease who require a primary total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Subject has hip disease that requires a total hip arthroplasty.
* Subject is willing to consent to participation in the study.
* Subject plans to be available for follow-up through study duration.
* Subject is of stable health and is free of or treated and stabilized for any condition that would prose excessive operating risk.

Exclusion Criteria:

* Subject has insufficient femoral bone stock.
* Subject has had major non-arthroscopic surgery to the study hip.
* Subject has physical, emotional or neurological conditions that would compromise the subjects compliance with postoperative rehabilitation and follow-up.
* Subject has a known sensitivity to materials in the device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The purpose of the current investigation is to compare migration of the device after implantation with a modular, short hip stem called the "MIS Stem" or a standard THA using the Synergy Hip System using RSA. The intended use of this product is for patients with inflammatory and non-inflammatory degenerative joint disease who require a primary total hip replacement.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2009-06-30 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard McCalden, MD, Principal Investigator — London Health Science Center; Beate Hanson, MD, PhD, Study Chair — Vice President, Global Clinical Strategy and Global Clinical Operations
Locations (1):
- London Health Sciences Center- University Hospital, London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled by 1 investigator in Canada. The study period was from 30 Jun 2009 to 22 Apr 2016.
Pre-assignment Details: Preoperative evaluation was conducted following signing of the ICF but prior to randomization. A total of 41 subjects had surgery for either MIS Stem or Synergy implantation.
Units Other Than Participants: hips
Groups:
- MIS Femoral Neck Stem: Designed to minimize the removal of bone from the femoral canal and the proximal neck. Along with a shortened length, the femoral stem uses a modular neck that allows for optimizing the offset angle to allow customization during surgery to better fit each patient. The modular neck features a standard taper consistent with various head options.
- Synergy Hip System: Standard total hip arthroplasty (THA) using total hip system.
Period: Overall Study
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Started | 21; 21 hips | 20; 20 hips
Completed | 18; 18 hips | 13; 13 hips
Not Completed | 3; 3 hips | 7; 7 hips
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Revision due to femoral stem loosening | 1 | 0
Not completed — Revision due to dislocation | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: 43 hips were randomized into the study, with 2 hips excluded, resulting in a total of 41 hips (4 bilateral hips) enrolled in the study - 20 Synergy hips and 21 MIS Stem hips
Groups:
- Total: Total of all reporting groups
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (7.93) | 65.8 (10.84) | 64.4 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 20 | 41
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 171.4 (9.12) | 168.5 (9.19) | 170.0 (9.16)
Weight [Mean (Standard Deviation); unit: kg] | 90.0 (18.22) | 88.0 (23.60) | 89.0 (20.78)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.7 (6.25) | 30.9 (7.34) | 30.8 (6.72)
Primary Diagnosis: Charnley Classification [Count of Participants; unit: Participants]
  Avascular necrosis: A unilateral hip joint disease | 1 | 0 | 1
  Osteoarthritis: A unilateral joint disease | 8 | 7 | 15
  Osteoarthritis: B1 bilateral hip joint disease | 9 | 10 | 19
  Osteoarthritis: C1 multi-joint arthroplasties | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Migration of the MIS Femoral Neck Stem Compared to the Synergy Hip System Using RSA (Translational Movement)
Description: Migration, or micromovement of the implant, was measured using RSA to compare the modular, short hip stem called the MIS Stem against a standard THA using Synergy Hip System.
Time Frame: Discharge (baseline), 6 weeks, 3 and 6 months, 1 and 2 years postoperative, change from baseline at 2 years reported
Population: Statistical comparisons were done using data from hips with all with RSA information at 2 years (20 MIS and 18 Synergy).
Measure: Mean (Full Range); unit: mm
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 20 | 18
mm
  Mean translation: Medial-lateral | 0.204 [-0.457 to 1.36] | 0.224 [-0.158 to 0.975]
  Mean translation: Proximal-distal | -0.942 [-5.86 to 0.026] | -0.322 [-1.57 to 0.281]
  Mean translation: Anterior-posterior | -0.031 [-1.05 to 1.00] | -0.328 [-2.44 to 0.692]
  Mean translation: Total three-dimensional | 1.090 [0.063 to 6.11] | 0.728 [0.175 to 3.06]

2. Secondary Outcome: Preoperative Total Harris Hip Score (HHS)
Description: The HHS is a physician tool to measure how a subject is doing after their hip was replaced. The HHS had a total range of 0-100 points and consisted of categories to assess Pain, Function, Absence of Deformity, Range of Motion, and Total Score. Each category was summarized and stratified into scores of Excellent (90-100), Good (80-89), Fair (70-79), Poor (60-69), and Very Poor (<60). Higher scores delineated better results for the subject.
Time Frame: Preoperative
Population: Data from hips with all with RSA information at pre-operative visit (21 MIS and 20 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 21 | 20
Participants
  Excellent (90-100) | 0 | 0
  Good (80-89) | 1 | 0
  Fair (70-79) | 1 | 1
  Poor (60-69) | 3 | 1
  Very Poor (<60) | 16 | 18

3. Secondary Outcome: 3 Months Postoperative Total Harris Hip Score (HHS)
Description: as for outcome 2
Time Frame: 3 months postoperative
Population: Data from hips with all with RSA information at 3 months (19 MIS and 16 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 19 | 16
Participants
  Excellent (90-100) | 10 | 7
  Good (80-89) | 6 | 6
  Fair (70-79) | 3 | 1
  Poor (60-69) | 0 | 2
  Very Poor (<60) | 0 | 0

4. Secondary Outcome: 1 Year Postoperative Total Harris Hip Score (HHS)
Description: as for outcome 2
Time Frame: 1 year postoperative
Population: Data from hips with all with RSA information at 1 year (21 MIS and 15 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 21 | 15
Participants
  Excellent (90-100) | 15 | 10
  Good (80-89) | 6 | 2
  Fair (70-79) | 0 | 2
  Poor (60-69) | 0 | 1
  Very Poor (<60) | 0 | 0

5. Secondary Outcome: 2 Years Postoperative Total Harris Hip Score (HHS)
Description: as for outcome 2
Time Frame: 2 years postoperative
Population: Data from hips with all with RSA information at 2 years (21 MIS and 16 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 21 | 16
Participants
  Excellent (90-100) | 14 | 7
  Good (80-89) | 4 | 6
  Fair (70-79) | 2 | 3
  Poor (60-69) | 0 | 0
  Very Poor (<60) | 1 | 0

6. Secondary Outcome: 3 Years Postoperative Total Harris Hip Score (HHS)
Description: as for outcome 2
Time Frame: 3 years postoperative
Population: Data from hips with all with RSA information at 3 years (15 MIS and 13 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 15 | 13
Participants
  Excellent (90-100) | 12 | 9
  Good (80-89) | 2 | 1
  Fair (70-79) | 0 | 2
  Poor (60-69) | 0 | 1
  Very Poor (<60) | 1 | 0

7. Secondary Outcome: 5 Years Postoperative Total Harris Hip Score (HHS)
Description: as for outcome 2
Time Frame: 5 years postoperative
Population: Data from hips with all with RSA information at 5 years (17 MIS and 12 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 17 | 12
Participants
  Excellent (90-100) | 9 | 8
  Good (80-89) | 4 | 3
  Fair (70-79) | 3 | 0
  Poor (60-69) | 0 | 1
  Very Poor (<60) | 1 | 0

8. Secondary Outcome: Preoperative Hip Disability Osteoarthritis Outcome Score (HOOS)
Description: The HOOS was a questionnaire that the subject completed focusing on hip pain, stiffness, and function relating to osteoarthritis of the hip. The HOOS consisted of 40 items assessing 5 subscales; Symptoms and Stiffness, Pain, Function of Daily Living, Function in Sport and Recreation, and hip-related Quality of Life.
  Pain included 10 items with a total score of 40 points Symptoms included 5 items with a total score of 20 points Function of Daily Living included 17 items with a total score of 68 points Function in Sport and Recreation included 4 items with a total score of 16 points Hip-related Quality of Life included 4 items with a total score of 16 points
  Each subscore was transformed into a worst-to-best scale (0-100), where 100 indicated no symptoms and 0 indicated extreme symptoms.
Time Frame: Preoperative
Population: Data from hips with all with RSA information at pre-operative visit (21 MIS and 20 Synergy).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 21 | 20
score on a scale
  Symptoms and Stiffness (0-100) | 47.4 (17.58) | 40.5 (16.05)
  Pain (0-100) | 37.1 (17.73) | 33.5 (17.44)
  Daily Living (0-100) | 41.0 (19.52) | 33.4 (16.97)
  Sports/ Recreational Activities (0-100) | 27.1 (19.70) | 22.8 (15.08)
  Quality of Life (0-100) | 23.2 (14.27) | 23.4 (13.43)

9. Secondary Outcome: 3 Months Postoperative Hip Disability Osteoarthritis Outcome Score (HOOS)
Description: as for outcome 8
Time Frame: 3 months postoperative
Population: Data from hips with all with RSA information at 3 months (19 MIS and 16 Synergy).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 19 | 16
score on a scale
  Symptoms and Stiffness (0-100) | 81.8 (9.75) | 77.2 (17.41)
  Pain (0-100) | 85.1 (12.40) | 76.9 (18.59)
  Daily Living (0-100) | 81.9 (11.63) | 76.0 (18.51)
  Sports/ Recreational Activities (0-100) | 67.4 (17.87) | 61.3 (20.82)
  Quality of Life (0-100) | 67.1 (17.03) | 66.0 (20.02)

10. Secondary Outcome: 1 Year Postoperative Hip Disability Osteoarthritis Outcome Score (HOOS)
Description: as for outcome 8
Time Frame: 1 year postoperative
Population: Data from hips with all with RSA information at 1 year (21 MIS and 15 Synergy).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 21 | 15
score on a scale
  Symptoms and Stiffness (0-100) | 87.9 (11.68) | 81.0 (13.39)
  Pain (0-100) | 85.0 (11.54) | 80.8 (17.52)
  Daily Living (0-100) | 85.1 (11.44) | 76.0 (18.77)
  Sports/ Recreational Activities (0-100) | 77.1 (19.09) | 66.3 (26.60)
  Quality of Life (0-100) | 76.2 (18.39) | 72.5 (18.87)

11. Secondary Outcome: 2 Years Postoperative Hip Disability Osteoarthritis Outcome Score (HOOS)
Description: as for outcome 8
Time Frame: 2 years postoperative
Population: Data from hips with all with RSA information at 2 years (21 MIS and 16 Synergy).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 21 | 16
score on a scale
  Symptoms and Stiffness (0-100) | 87.9 (11.57) | 82.2 (12.11)
  Pain (0-100) | 84.2 (15.80) | 81.7 (21.09)
  Daily Living (0-100) | 82.4 (17.61) | 72.1 (22.41)
  Sports/ Recreational Activities (0-100) | 76.8 (20.46) | 74.6 (23.88)
  Quality of Life (0-100) | 83.3 (20.57) | 75.4 (16.84)

12. Secondary Outcome: 3 Years Postoperative Hip Disability Osteoarthritis Outcome Score (HOOS)
Description: as for outcome 8
Time Frame: 3 years postoperative
Population: Data from hips with all with RSA information at 3 years (15 MIS and 13 Synergy).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 15 | 13
score on a scale
  Symptoms and Stiffness (0-100) | 88.0 (17.91) | 81.9 (17.26)
  Pain (0-100) | 84.0 (18.51) | 85.8 (17.45)
  Daily Living (0-100) | 86.0 (19.38) | 73.0 (23.15)
  Sports/ Recreational Activities (0-100) | 77.9 (22.76) | 75.0 (19.93)
  Quality of Life (0-100) | 82.1 (22.39) | 79.8 (25.91)

13. Secondary Outcome: 5 Years Postoperative Hip Disability Osteoarthritis Outcome Score (HOOS)
Description: as for outcome 8
Time Frame: 5 years postoperative
Population: Data from hips with all with RSA information at 3 years (17 MIS and 12 Synergy).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 17 | 12
score on a scale
  Symptoms and Stiffness (0-100) | 85.3 (15.96) | 84.4 (20.12)
  Pain (0-100) | 81.2 (18.95) | 78.1 (25.45)
  Daily Living (0-100) | 76.7 (21.51) | 71.0 (25.33)
  Sports/ Recreational Activities (0-100) | 68.4 (30.09) | 50.0 (45.54)
  Quality of Life (0-100) | 71.0 (28.38) | 75.0 (29.07)

14. Secondary Outcome: Preoperative Radiographic Assessments
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: Preoperative
Population: Data from all enrolled hips who received a study device (21 MIS and 20 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 21 | 20
Participants
  No Problems on Checklist: Yes | 21 | 20
  No Problems on Checklist: No | 0 | 0
  Acetabular Cup Subsidence: Yes | 0 | 0
  Acetabular Cup Subsidence: No | 21 | 20
  Stem Subsidence: Yes | 0 | 0
  Stem Subsidence: No | 21 | 20
  Evidence of Acetabular Component Failure: Yes | 0 | 0
  Evidence of Acetabular Component Failure: No | 21 | 20
  Evidence of Femoral Component Failure: Yes | 0 | 0
  Evidence of Femoral Component Failure: No | 21 | 20

15. Secondary Outcome: 3 Months Postoperative Radiographic Assessments
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 3 months postoperative
Population: Data from hips with all with RSA information at 3 months (19 MIS and 16 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 19 | 16
Participants
  No Problems on Checklist: Yes | 19 | 16
  No Problems on Checklist: No | 0 | 0
  Acetabular Cup Subsidence: Yes | 0 | 0
  Acetabular Cup Subsidence: No | 19 | 16
  Stem Subsidence: Yes | 0 | 0
  Stem Subsidence: No | 19 | 16
  Evidence of Acetabular Component Failure: Yes | 0 | 0
  Evidence of Acetabular Component Failure: No | 19 | 16
  Evidence of Femoral Component Failure: Yes | 0 | 0
  Evidence of Femoral Component Failure: No | 19 | 16

16. Secondary Outcome: 1 Year Postoperative Radiographic Assessments
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 1 year postoperative
Population: Data from hips with all with RSA information at 1 year (20 MIS and 15 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 20 | 15
Participants
  No Problems on Checklist: Yes | 15 | 11
  No Problems on Checklist: No | 5 | 4
  Acetabular Cup Subsidence: Yes | 0 | 0
  Acetabular Cup Subsidence: No | 20 | 15
  Stem Subsidence: Yes | 0 | 0
  Stem Subsidence: No | 20 | 15
  Evidence of Acetabular Component Failure: Yes | 0 | 0
  Evidence of Acetabular Component Failure: No | 20 | 15
  Evidence of Femoral Component Failure: Yes | 0 | 0
  Evidence of Femoral Component Failure: No | 20 | 15

17. Secondary Outcome: 2 Years Postoperative Radiographic Assessments
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 2 years postoperative
Population: Data from hips with all with RSA information at 2 years (21 MIS and 16 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 21 | 16
Participants
  No Problems on Checklist: Yes | 11 | 12
  No Problems on Checklist: No | 10 | 4
  Acetabular Cup Subsidence: Yes | 0 | 0
  Acetabular Cup Subsidence: No | 21 | 16
  Stem Subsidence: Yes | 1 | 0
  Stem Subsidence: No | 20 | 16
  Evidence of Acetabular Component Failure: Yes | 0 | 0
  Evidence of Acetabular Component Failure: No | 21 | 16
  Evidence of Femoral Component Failure: Yes | 0 | 0
  Evidence of Femoral Component Failure: No | 21 | 16

18. Secondary Outcome: 3 Years Postoperative Radiographic Assessments
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 3 years postoperative
Population: Data from all enrolled hips who received a study device (15 MIS and 13 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 15 | 13
Participants
  No Problems on Checklist: Yes | 8 | 7
  No Problems on Checklist: No | 7 | 6
  Acetabular Cup Subsidence: Yes | 0 | 0
  Acetabular Cup Subsidence: No | 15 | 13
  Stem Subsidence: Yes | 0 | 0
  Stem Subsidence: No | 15 | 13
  Evidence of Acetabular Component Failure: Yes | 0 | 0
  Evidence of Acetabular Component Failure: No | 15 | 13
  Evidence of Femoral Component Failure: Yes | 0 | 0
  Evidence of Femoral Component Failure: No | 15 | 13

19. Secondary Outcome: 5 Years Postoperative Radiographic Assessments
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 5 years postoperative
Population: Data from all enrolled hips who received a study device (17 MIS and 12 Synergy).
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 17 | 12
Participants
  No Problems on Checklist: Yes | 13 | 11
  No Problems on Checklist: No | 4 | 1
  Acetabular Cup Subsidence: Yes | 0 | 0
  Acetabular Cup Subsidence: No | 17 | 12
  Stem Subsidence: Yes | 0 | 0
  Stem Subsidence: No | 17 | 12
  Evidence of Acetabular Component Failure: Yes | 0 | 0
  Evidence of Acetabular Component Failure: No | 17 | 12
  Evidence of Femoral Component Failure: Yes | 0 | 0
  Evidence of Femoral Component Failure: No | 17 | 12

20. Primary Outcome: Migration of the MIS Femoral Neck Stem Compared to the Synergy Hip System Using RSA (Rotational Movement)
Description: as for outcome 1
Time Frame: Discharge (baseline), 6 weeks, 3 and 6 months, 1 and 2 years postoperative, change from baseline at 2 years reported
Population: Statistical comparisons were done using data from hips with all with RSA information at 2 years (20 MIS and 18 Synergy).
Measure: Mean (Full Range); unit: degrees
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
Number analyzed (Participants) | 20 | 18
degrees
  Mean rotation: Anterior-posterior | -0.475 [-2.70 to 0.19] | -0.006 [-0.74 to 0.92]
  Mean rotation: Internal-external | 0.958 [-0.43 to 5.69] | 1.414 [-0.71 to 11.65]
  Mean rotation: Varus-valgus tilt | -0.463 [-2.79 to 0.21] | -0.091 [-1.29 to 0.17]

ADVERSE EVENTS:
Time Frame: From signed consent to the completion of the study at the 5-year follow-up visit, or early termination/subject withdrawal, whichever came first.
Arm/Group | MIS Femoral Neck Stem | Synergy Hip System
All-Cause Mortality (participants affected / at risk) | 0/21 | 1/20
Serious Adverse Events (participants affected / at risk) | 2/21 | 4/20
Other Adverse Events (participants affected / at risk) | 15/21 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIS Femoral Neck Stem (N=21) | Synergy Hip System (N=20)
Loose femoral stem (Product Issues) | 1 (1) | 0 (0)
Subluxed patella/medial patellar retinacular repair (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis total knee replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adverse soft tissue reaction secondary to dual taper from modular neck (Product Issues) | 1 (1) | 0 (0)
Stroke (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hip dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Hip instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Unresectable pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIS Femoral Neck Stem (N=21) | Synergy Hip System (N=20)
Superficial wound infection (Infections and infestations) | 1 (1) | 0 (0)
Leg Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Torn meniscus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (8) | 6 (9)
Degenerative changes with narrowing of the joint line and osteophytic changes (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radiographic review finding of 5mm stem subsidence from fibrous ingrowth hip stem (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stem revision right hip replacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Bleeding duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subphrenic abscess (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stitch abscess (Infections and infestations) | 1 (1) | 1 (1)
Femoral hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Medial compartmental arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Reaction to metal debris/ metal allergy (Product Issues) | 1 (1) | 0 (0)
Pain in study hip (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Partial peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Buttock pain/soreness/discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stress shielding as indicated on radiographic findings CRF (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Lysis over greater trochanter of total hip replacement (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain in anterior aspect of knee possible flare-up of scar tissue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hip dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Fractured ankle (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
L2-3,L4-5 Spinal stenosis;L5-S1 right-sided lateral recess stenosis, iatrogenic dural tear L4-5 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Greater trochanteric pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nonoperative tibial plateau fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There was a decreased compliance rate at the 3-year follow-up visit and an increased termination rate by the 5-year follow-up visit resulting in smaller sample sizes for data collection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less